CLINICAL TRIAL: NCT04057963
Title: The Inspiratory Muscle Training in Patients With Non-Specific Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gamze YALCINKAYA, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3758-GOA
Record Dates: First submitted 2019-08-11; First posted 2019-08-15 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Neck Pain
Keywords: Inspiratory Muscle Training; Exercise; Cervical Posture
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional plus Functional Inspiratory Muscle Training Group (Experimental): Conventional program plus functional inspiratory muscle training will be carried out three sessions per week during the six weeks. The content of the program will be the same as for the conventional group. Additional functional inspiratory muscle training will be began with 50% of the maximal inspiratory pressure value in a specific device and it will be progressed 5% every week according to the tolerance.
  Interventions: Other: Conventional plus Functional Inspiratory Muscle Training Group
- Conventional Physiotherapy Program (Active Comparator): Conventional program will be carried out three sessions per week during the six weeks. Cervical mobilization techniques (glidings-grade 2) of cyriax will be applied in the direction of lateral flexion and rotation. Stretching exercises, craniovertebral flexion exercise and scapulothoracic strengthening exercises will be performed.
  Interventions: Other: Conventional Physiotherapy Program

INTERVENTIONS:
Other: Conventional plus Functional Inspiratory Muscle Training Group — functional inspiratory muscle training is an exercise program that practises gradual training of the diaphragm muscle.
  Arms: Conventional plus Functional Inspiratory Muscle Training Group
Other: Conventional Physiotherapy Program — conventional physiotherapy is a treatment program consisting of evidence based modalities as mobilization and specific exercises.
  Arms: Conventional Physiotherapy Program

SUMMARY:
The aim of the present study is to investigate the effects of additional functional inspiratory muscle training in individuals with non-specific chronic neck pain.

DETAILED DESCRIPTION:
Patients participating in the study will be divided two parallel groups. The patients in study group will instruct to perform both functional inspiratory muscle training and conventional treatments for neck pain, the patients in the control group will instruct to perform just conventional treatments. The severity of the pain, disability, fear of movement and depression levels will be assessed by visual analog scale, neck disability index, Tampa Scale of kinesiophobia and beck depression inventory, respectively. Neck postures (craniovertebral angle) will be evaluated by photogrammetric method.Endurance of deep cervical flexor muscles will be measured using Stabilizer Pressure Biofeedback Unit with cranio-cervical flexion test. Pain threshold will be measured by algometer from the middle point of upper trapezius. Cervical proprioceptions will be evaluated by laser pointer method in the right and left rotational directions. In addition, diaphragma thickness will be measured by two-dimensional ultrasonography. Assessments were repeated before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* NDI score above 15
* Be able to adapt exercise commands
* Neck pain for at least six months
* Agree to participate in the study

Exclusion Criteria:

History of spinal surgery Traumatic cervical injuries Acute or chronic musculoskeletal pain other than neck pain Serious comorbidities (neurological, neuromuscular, cardiological, psychiatric) Tumoral conditions Obesity (Body Mass Index-BMI> 40)

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-10 (Actual); Primary Completion 2021-08-10 (Estimated); Study Completion 2021-08-10 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain Severity | change from baseline in pain severity at 6 weeks
  Patients' resting pain intensities will be assessed by Visual Analog Scale. (a 10 cm horizontal line). There is two anchors in the tips of the visual analog scale and while the zero represented "no pain", ten indicated "excessive pain". The length from the zero to marked point was recorded in cm.
Changes in Disability | change from baseline in disability at 6 weeks
  Patients' disability levels will be assessed by neck disability index. The questionnaire has ten sections; pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each item is scored between zero (no disability) and five (total disability). The maximum score is therefore 50. Higher scores indicates having more disability.
Changes in Fear of Movement | change from baseline in disability at 6 weeks
  Patients' fear of movement will be assesed by Tampa Kinesiophobia Scale. The scale has 17 pain statements, and the patient selected her agreement for each question using a 4-point scale. The maximum score is 68. Higher score indicates having more fear of movement.
Changes in Depression | change from baseline in disability at 6 weeks
  Patients' depression levels will be assessed by Beck Depression Inventory. composed 21 questions. The maximum total score is 63. Higher scores demonstrate greater level of depression

SECONDARY OUTCOMES:
Craniovertebral Angle | change from baseline in disability at 6 weeks
  Photogrammetric method will be used to evaluate craniovertebral angle.
Pain threshold | change from baseline in disability at 6 weeks
  Pain threshold will be measured by Algometer device.
Cervical Proprioception | change from baseline in disability at 6 weeks
  Cervical Proprioception will be evaluated by laser pointer method.
Cranio-cervical flexion endurance | change from baseline in disability at 6 weeks
  Cranio-cervical flexion endurance (activation score) will be measured by stabilizer pressure biofeedback unit.
Diaphragma thickness | change from baseline in disability at 6 weeks
  Diaphragma thickness will be measured by two dimensional ultasonography
Respiratory Muscle Strength | change from baseline in disability at 6 weeks
  Respiratory Muscle Strength (maximum inspiratory and expiratory mouth pressure) will be measured by Micro RPM device

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Dokuz Eylul University, Department of Neurosurgery, Izmir, Inciraltı
  - Dokuz Eylul University, School of Physical Therapy and Rehabilitation, Izmir

IPD SHARING:
Plan to Share IPD: Undecided